CLINICAL TRIAL: NCT06580197
Title: Application of Auricular Acupuncture Therapy Based on Real-World Studies After Abdominal Surgery
Brief Title: The Role of AAT After Abdominal Surgery Based on RWS
Status: Recruiting | Type: Observational
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: K6357
Record Dates: First submitted 2024-08-28; First posted 2024-08-30 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-08

CONDITIONS: Acupuncture, Ear; Gastroparesis
MeSH Terms: conditions — Gastroparesis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Surgical control group (Group A): Patients who received ear acupuncture treatment (≥ 1 time) due to perioperative anxiety, pain, prevention/treatment of DGF, or other indications for ear acupuncture treatment in actual diagnosis and treatment were divided into two groups based on exposure factors. Patients who received ear acupuncture treatment were included in the surgical observation group (Group B), while other patients were included in the surgical control group (Group A). Both groups of patients were from the basic surgical ward of Peking Union Medical College Hospital and were planning to undergo abdominal surgeries such as Whipple, pancreaticoidectomy, and subtotal gastrectomy;
- Surgical observation group (Group B): Patients who received ear acupuncture treatment (≥ 1 time) due to perioperative anxiety, pain, prevention/treatment of DGF, or other indications for ear acupuncture treatment in actual diagnosis and treatment were divided into two groups based on exposure factors. Patients who received ear acupuncture treatment were included in the surgical observation group (Group B), while other patients were included in the surgical control group (Group A). Both groups of patients were from the basic surgical ward of Peking Union Medical College Hospital and were planning to undergo abdominal surgeries such as Whipple, pancreaticoidectomy, and subtotal gastrectomy;
  Interventions: Other: Auricular Acupoint Therapy
- Healthy control group (Group C): According to the surgical observation group (Group B), the healthy control group (Group C) consisted of healthy volunteers from the same period at the Beijing Union Medical College Hospital Health Examination Center.

INTERVENTIONS:
Other: Auricular Acupoint Therapy — Ear point diagnosis and treatment is one of acupuncture and moxibustion methods, which originates from the theory of acupuncture and moxibustion meridians and is the product of the combination of modern Chinese medicine and western medicine, including two parts: auricular acupoint diagnosis and auriculotherapy. Ear point diagnosis refers to the determination of auricle positive reaction points through vision, touch, pressure and other methods to diagnose diseases in some parts of the body on the basis of ear point theory. Ear point treatment refers to the use of certain therapeutic devices on ear points to achieve the purpose of prevention and treatment of diseases by stimulating ear points, which are often carried out simultaneously in clinical practice.
  Groups: Surgical observation group (Group B)

SUMMARY:
Delayed gastric emptying (DGE) after surgery mainly occurs after gastrointestinal surgery A functional gastric emptying disorder, clinically characterized by weak or absent gastric peristalsis, gastric motility disorders, or gastric emptying Gastric retention, fullness, nausea and other uncomfortable symptoms caused by delay.This study is based on clinical diagnosis and treatment practice, observing, collecting, and analyzing Whipple surgery, pancreatectomy, and gastric cancer Perioperative data of subtotal resection surgery, mainly observing the diagnosis and treatment of ear acupoints in Whipple surgery, pancreatectomy, and subtotal gastrectomy.The application effect of DGE after resection surgery, exploring the diagnosis and treatment of ear acupoints in Whipple surgery, pancreatic body and tail resection surgery, and Diagnostic value of perioperative related diseases in abdominal surgery such as subtotal gastrectomy, and collection of health records.By comparing and analyzing the ear acupoint information of patients with abdominal tumors, we aim to explore the ear acupoints of the volunteers. The possible relationship between image and resistance specificity and common tumors in the abdominal cavity.

ELIGIBILITY:
Inclusion Criteria:

- 1) Age range: 40-70 years old (40 ≤ y ≤ 70), gender is not limited. 2) Accept abdominal surgeries including Whipple's surgery, pancreatectomy, and subtotal gastrectomy.

3) The subjects/guardians are able to understand the purpose of the trial, demonstrate sufficient compliance with the trial protocol, and sign an informed consent form (ICF)

Exclusion Criteria:

* 1) Severe postoperative complications such as heart disease, pulmonary embolism, cerebral infarction, abdominal infection, and abdominal bleeding; 2) Patients with organic changes such as adhesions and obstructions indicated by imaging examinations such as gastrointestinal imaging; 3) The patient has damage, redness, bleeding, infection, and other conditions in both ears that are not suitable for ear acupuncture treatment.

Inclusion and exclusion criteria for the health group

Inclusion Criteria:

1. Age range: 40-70 years old (40 ≤ y ≤ 70), gender is not limited.
2. No history of abdominal surgery or tumor, and no significant abnormalities were found through abdominal imaging examination.
3. The subjects/guardians are able to understand the purpose of the trial, demonstrate sufficient compliance with the trial protocol, and sign an informed consent form (ICF).

Exclusion Criteria:

1. Symptoms of digestive discomfort such as diarrhea, constipation, and vomiting have been present for the past 30 days.
2. The patient has conditions such as damage, redness, bleeding, and infection in both ears that affect the assessment of ear acupoint information.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Research subjects: Surgical group: (1) Patients who were scheduled to undergo abdominal surgeries such as Whipple, pancreatectomy, and subtotal gastrectomy at Peking Union Medical College Hospital from June 2024 to June 2026.
  Health group: (2) Patients who visited the Health Examination Center of Peking Union Medical College Hospital from June 2024 to June 2026.
Sampling Method: Non-Probability Sample
Enrollment: 159 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Clinical total effective rate | On the third day after surgery
  The clinical total effective rate of ear acupuncture treatment for postoperative DGE in the abdomen, including Whipple surgery, pancreatectomy, and subtotal gastrectomy.
  Efficacy evaluation criteria: Measure the subjective symptom score (Gastroparesis Cardinal Symptom Index, GCSI score) of patients with gastroparesis on the third day after surgery, and calculate the clinical efficacy index of ear acupuncture treatment using the following formula (efficacy index=[(total score of symptoms before treatment - total score of symptoms after treatment) ÷ total score of symptoms before treatment × 100%]). Among them, significant effect: efficacy index>75%; Effective: Efficacy index of 25% to 75%; Invalid: Efficacy index<25%. Total effective rate=(number of significantly effective cases+number of effective cases)/total number of cases x 100%.
Perioperative Anxiety Scale-7 (PAS-7) | 24±2h after the start of AP or first visit, 12±2h before surgery, and 2 h before surgery
  This scale was used to evaluate the anxiety of patients before surgery. This scale evaluates some of the patient's conditions regarding the operation, and then, based on the actual situation during the days of hospitalization, selects the appropriate option among 5 options, circling the corresponding numbers. The higher the score, the more severe the patient's preoperative anxiety level.

SECONDARY OUTCOMES:
Modified Pittsburgh Sleep Quality Index (M-PSQI) | 24±2h after the start of AP or first visit (T1), 12±2h before surgery (T2), and 72±2h post-operatively
  To accommodate the short treatment duration and unique ward environment of hospitalized patients, this study modified the Pittsburgh Sleep Quality Index (PSQI) to develop an adapted version (M-PSQI) for short-term sleep assessment. The scale consists of 24 items (19 self-rated + 5 caregiver-rated), with scoring based on the 19 self-rated items, which assess the following dimensions:
  1. Sleep Process Metrics: Sleep latency, total sleep duration, wake time
  2. Sleep Disturbance Manifestations: Difficulty falling asleep, nocturnal awakening frequency, environmental/physiological sleep disruptions
  3. Subjective Sleep Quality: Patients' overall evaluation of sleep quality
  4. Medication Use: Frequency of sedative-hypnotic drug use
  5. Daytime Functional Impairment: Difficulty maintaining wakefulness, reduced task performance efficiency The scale adopts a 7-factor structure, with each factor scored on a 0-3 scale. The total score ranges from 0 to 21, with higher scores indicating more severe sleep
Self-Rating Anxiety Scale (SAS) Score | Multiple time points before and after surgery
  The Self-Rating Anxiety Scale (SAS) was used to comprehensively evaluate the baseline anxiety levels of patients undergoing total knee arthroplasty (TKA) before surgery.
  Key Features of the SAS:
  Assessment Period: The scale assesses the patient's anxiety levels over the past week.
  Scoring Method: Forward-scoring items: Responses A, B, C, and D are scored as 1, 2, 3, and 4 points, respectively. Reverse-scoring items: Responses are scored as 4, 3, 2, and 1 points, respectively. The reverse-scored items are 5, 9, 13, 17, and 19 (highlighted in bold in the table below).All other items are forward-scored.
  Score Calculation and Interpretation: The raw score is obtained by summing the scores of all 20 items. The raw score is then multiplied by 1.25 and rounded to the nearest whole number to derive the standard score. The cutoff value for anxiety is 50. Higher scores indicate more pronounced anxiety tendencies.
  50-59: Mild anxiety 60-69: Moderate anxiety 70 and above: Severe anxiety.
Patient Satisfaction with Pre-operative Preparation Assessed with the Visual Analogue Scale (VAS-Satisfaction) | Preoperative
  The Visual Analogue Scale for Satisfaction (VAS-Satisfaction) is a simple, validated tool used to measure a patient's subjective satisfaction with their pre-operative preparation. It consists of a 100-mm horizontal line anchored by two extreme statements: Left anchor (0 mm): "Not satisfied at all"; Right anchor (100 mm): "Completely satisfied".
  The patient marks a point on the line corresponding to their level of satisfaction with the pre-operative process (This includes the information provided before surgery, the attitude of the medical staff, the arrangement of the preoperative process, and the overall experience of preoperative preparation). The score is quantified by measuring the distance (in mm) from the left anchor to the patient's mark, yielding a numerical value between 0 (lowest satisfaction) and 100 (highest satisfaction).
Visual Analogue Scale for Pain (VAS-Pain) | Multiple time points after surgery
  The Visual Analogue Pain Score (VAS-Pain) is a tool used to quantify a patient's subjective pain intensity using a straight line of 100 millimeters (10 cm) with two ends representing "no pain" and "most severe pain", and the patient assesses their pain level by marking their position on the straight line.

CONTACTS AND LOCATIONS:
Overall Officials: weibin Wang, Principal Investigator — Peking Union Medical College Hospital (CAMS)
Locations (1):
- Peking union medical college hospital, Beijing, Beijing Municipality, China